CLINICAL TRIAL: NCT00767494
Title: Travoprost/Brinzolamide Fixed Combination Versus Travatan and Versus AZOPT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Project Cancelled
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-07-63
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2009-07

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: OAG; OH; Open-angle glaucoma or ocular hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Glaucoma, Open-Angle | interventions — Travoprost; brinzolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Travoprost/Brinzolamide AM, Vehicle PM
  Interventions: Drug: Travoprost/Brinzolamide fixed combination
- 2 (Experimental): Travoprost/Brinzolamide PM, Vehicle AM
  Interventions: Drug: Travoprost/Brinzolamide fixed combination
- 3 (Active Comparator): AZOPT AM and PM
  Interventions: Drug: Azopt
- 4 (Active Comparator): TRAVATAN PM, Vehicle AM
  Interventions: Drug: Travatan

INTERVENTIONS:
Drug: Travoprost/Brinzolamide fixed combination — Eye Drops, suspension once daily
  Arms: 1; 2
Drug: Azopt — Eye Drop Suspension, 1 drop BID
  Arms: 3
Drug: Travatan — Eye Drop Solution, 1 drop BID
  Arms: 4

SUMMARY:
The purpose of the study is to compare the IOP lowering efficacy of Travoprost/Brinzolamide dosed daily in the morning or evening, vs TRAVATAN dosed once daily in the evening, and vs. AZOPT dosed BID in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 YOA or older
* Either gender or any race
* OAG or OHT
* Currently on stable (at least 4 weeks) IOP lowering medication
* IOP at screening visit â‰¥ 18mmHg in at least one eye
* Mean IOP in same eye (at both eligibility 1&2 visits
* 24 and 36 mmHg at 9AM
* 21 and 36 mmHg at 11AM and 4PM
* Able to discontinue use of IOP lowering medication for a minimum wash out period of 5 to 28 days prior to eligibility visit 1

Exclusion Criteria:

Related to disease condition being investigated (OAG or OHT) in either eye

* Severe central visual field loss
* Angle shaffer grade < 2
* C/D ratio >0.8(horizontal or vertical measurement)

Related to ocular patient history or current ocular condition in either eye

* BSCVA worse than 55 ETDRS letters read (equivalent to approximately 20/80 Snellen or 0.25 decimal)
* Ocular infection or inflammation or laser surgery within the last 3 months
* Intraocular surgery or trauma with the last 6 months
* Any abnormality preventing reliable applanation tonometry
* History or chronic, recurrently or current severe inflammatory disease
* History of or current clinically significant or progressive retinal disease
* History of or current ocular pathology(including severe dry eye) that would affect the conduct of the study

Related to systemic or ocular medication in either eye

* Allergy/hypersensitivity to study medications
* Unable to discontinue glucocorticoid at least 4 weeks prior to the study or unable to remain off these medications during the study period
* Use of oral CAIs during the study
* Recent use (<4 weeks prior to the study) of Aspirin (>1 gram)
* Less than 30 days stable dosing regimen of medications used on a chronic basis that may affect IOP
* Therapy with another investigational agent within 30 days prior to the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Mean IOP | 9, 11, and 16:00 time points at Week 12

SECONDARY OUTCOMES:
Mean diurnal IOP at Week 12 | results pooled across 9,11, and 16:00 time points

CONTACTS AND LOCATIONS:
Locations (1):
- Brussels, Belgium